CLINICAL TRIAL: NCT05803538
Title: Participant Centered Active Surveillance for Adverse Event Following Measles Immunization in Gedeo Zone, Ethiopia, 2022. A Multi-center Open-label Randomized Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dilla University (Other)
Responsible Party: Principal Investigator, Dawit Getachew Getachew, Mr., Dilla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ETDU005
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Measles
Keywords: Participant Centered Active Surveillance; Adverse Event; Measles Immunization
MeSH Terms: conditions — Measles | interventions — Interviews as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SMS (Experimental)
  Interventions: Device: SMS, telephone interview or diary card
- Telephone interview (Experimental)
  Interventions: Device: SMS, telephone interview or diary card
- Diary card (Experimental)
  Interventions: Device: SMS, telephone interview or diary card
- Usual Care (Active Comparator)
  Interventions: Device: SMS, telephone interview or diary card

INTERVENTIONS:
Device: SMS, telephone interview or diary card — SMS, telephone interview or diary card

SUMMARY:
Introduction Participant centered active adverse event following immunization (AEFI) surveillance can offer real time vaccine safety data and help in signal detection. Evidence showed that it is still difficult to get AEFI from passive reporting in Ethiopia. Vast novel method of enhanced AEFI surveillance has been practiced globally. However, those methods had serious limitations including the requirement of high resource and expertise. Hence, there is a need to find the most flexible low cost and integrated AEFI surveillance system. To the best of our knowledge, there has no published research in Ethiopia which compare Participant diary, SMS, and telephone interview for the purpose of active AEFI surveillance.

Objective: To assess participant centered active adverse event surveillance following measles immunization at Gedeo Zone health facilities, Ethiopia.

Method: An open randomized trial will be employed from October 1, 2022- December 1, 2023, at Gedio Zone health facilities. All parents, care givers/guardians whose child receive vaccine during the study period in the study site will be included in the study. A total of 391participants will be randomized to SMS, telephone interview or diary card group using random number generator on Excel. Every participant will be contacted on day seven to request them whether they experience any AEFI. Differences in proportions will compared using chi-square tests. A 0.05 level of significance will be used for all analyses. Independent sample t-tests will be used to compare the mean time (in days) required to collect complete AEFI data by SMS, telephone interview and diary card. Multinominal logistic regression analyses will be used assess the factors associated with effective use of tailored SMS, telephone interview and diary card for the AEFI active surveillance. To further investigate the association between the vaccine and the adverse events and factors associated with vaccine binary and multi variable logistic regression will be used.

ELIGIBILITY:
Inclusion Criteria:

* Parents, care givers/guardians, whose child receive vaccine.
* ≥18 years of age.
* Willing to adhere to study procedures, which will include a randomization.
* Willing to participate

Exclusion Criteria:

* Unable to give informed consent because of cognitive impairment.
* Those who are both illiterate and don't have mobile phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 391 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Response rate | 7 days
  To compare response rate of tailored SMS, telephone interview and diary card for the AEFI active surveillance

SECONDARY OUTCOMES:
AEFI's reported from each group and feasibility of participant centered AEFI active surveillance | 7days

CONTACTS AND LOCATIONS:
Locations (1):
- Dilla University, Awasa, Snnpr, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Assefa DG, Tesefaye T, Bekele E, Geberemickeal G, Mebratu A, Ejigu AG, Nigatu T, Zeleke ED. Active surveillance of immunization adverse effects: a multicentre, open-label, three-arm randomized uncontrolled trial in Ethiopia. Int Health. 2025 Mar 4;17(2):195-204. doi: 10.1093/inthealth/ihae040. PMID 38828522